CLINICAL TRIAL: NCT02869698
Title: Spectral Dynamic Imaging of Cognitive Functions in Epileptic Patients Explored
Brief Title: Spectral Dynamic Imaging of Cognitive Functions in Epileptic Patients Explored Stereoelectroencephalography
Acronym: ISDETSEEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 38RC09.012
Record Dates: First submitted 2016-08-04; First posted 2016-08-17 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Evaluation of cognitive functions by Spectral Dynamic Imaging (Experimental): Evaluation of cognitive functions by SDI will be conducted during the exploration SEEG (which usually lasts from 1 to 3 weeks), and started a few days after implantation of intracranial electrodes
  Interventions: Procedure: Spectral Dynamic Imaging; Device: Hybride electrode; Device: Macro electrode

INTERVENTIONS:
Procedure: Spectral Dynamic Imaging
Device: Hybride electrode
  Other Names: AdTech Medical Instrument Corporation
Device: Macro electrode
  Other Names: DIXI Microtechniques

SUMMARY:
This prospective research aims to develop the use of Spectral Imaging in addition Dynamics of cortical electrical stimulation to identify major anatomical and functional networks in epileptic patients candidates for surgery and explored by stereoencephalography, to minimize risk of post-surgical cognitive deficits.

DETAILED DESCRIPTION:
Cognitive deficits after epilepsy surgery are poorly known particularly because the tools used to evaluate them. In addition, the prevention of certain postoperative deficits, is extremely difficult because of the lack of robust markers to anticipate. The various examinations conventionally used for this purpose (neuropsychological testing, functional MRI and cortical stimulation) does indeed provide insufficient information or difficult to interpret, so the development of improved methods appears as an imperative in the field of the epilepsy surgery.

SID appears as such particularly adapted to the case of epileptic patients explored SEEG to provide individualized cognitive map millimeter thereof without requiring, for additional invasive act, or risk of inducing unintended crisis. In practice, this clinical research project should lead to the definition of several simple cognitive tasks which, together, could be achieved by each volunteer patient in two or three hours, and then analyzed in a similar time to provide fast, even the patient is still explored SEEG and even before cortical electrical stimulation, a list of brain regions involved in most major cognitive functions.

ELIGIBILITY:
Inclusion Criteria:

* Drug-resistant partial epilepsy justifying a SEEG exploration
* Intellectual capacities compatible with the award of cognitive tasks

Exclusion Criteria:

* Pregnant or lactating women
* Patient deprived of liberty by a judicial or administrative
* Major patient subject to a measure of legal protection

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2009-06; Primary Completion 2017-05 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Functional brain mapping procedure using the EEG signal intracranial to minimize the risk of cognitive deficits associated with resection of the epileptogenic zone. | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Philippe KAHANE, Principal Investigator — University Hospital, Grenoble
Locations (2):
- France (2):
  - University Hospital Grenoble, Grenoble
  - University Hospital Lyon, Lyon

IPD SHARING:
Plan to Share IPD: No